CLINICAL TRIAL: NCT01430013
Title: Phase II Trial of Endostar Combined With CHOPT for T Cell Lymphoma
Brief Title: Trial of Endostar Combined With CHOPT for T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2367240
Record Dates: First submitted 2011-07-11; First posted 2011-09-07 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2011-09

CONDITIONS: T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — endostar protein; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endostar (Experimental): CHOPT chemotherapy plus Endostar
  Interventions: Drug: Endostar and CHOPT

INTERVENTIONS:
Drug: Endostar and CHOPT — Endostar 7.5mg/m2, for iv for continuous 14 days cyclophosphamide, pirarubicin, vincristine, teniposide, prednisone
  Other Names: Endostatin

SUMMARY:
To evaluate the efficacy and safety of Endostar combined with CHOPT in the treatment of T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 to 70 years old.
2. Diagnosis of T cell lymphoma according to WHO Classification, without antitumor therapy
3. At least 1 measurable tumor mass (greater than 1.5cm in the longest dimension and greater than 1.0 in the short axis)
4. Eastern Cooperative Oncology Group status 0-2
5. White blood cell≥4.0×109cells/L; Absolute neutrophil count (ANC) ≥1.5×109cells /L; Platelets≥100×109cells/L
6. Alanine transaminase (ALT) ≤2×upper limit of normal(ULN); Aspartate transaminase (AST) ≤2×ULN; Total Bilirubin≤1.5×ULN; Creatinine in normal range

Exclusion Criteria:

1. No active central nervous system lymphoma or brain tumor
2. Suppurative inflammation,Chronic infection
3. Severe heart disease, conclusion: congestive heart failure; uncontrolled cardiac arrhythmia; myocardial infarction; refractory hypertension
4. psychiatric history
5. Primary cutaneous T cell lymphoma
6. Pregnant or lactating women
7. Concurrent treatment with another investigational agent
8. Accept radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
efficacy including overall response rate, progression free survival and overall survival | 1 year
  According to International Workshop Criteria, the number of participants with complete remission, partial remission and stable disease as a measure of efficacy.progressive free survival and overall survival of the participants are the second measure of efficacy

SECONDARY OUTCOMES:
safety of Endostar combined with CHOPT chemotherapy | 1 year
  Number of participants with adverse events as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Huaqing wang, MD, Principal Investigator — Tianjin Medical University Cancer Institue and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China